CLINICAL TRIAL: NCT04613765
Title: A Mixed Method Study Design to Explore Adherence of Haematological Cancer Patients to Oral Anticancer Medication in a Multilingual and Multicultural Outpatient Setting: the MADESIO Protocol
Brief Title: A Mixed Method to Study Adherence to Oral Anticancer Medications in a Multilingual and Multicultural Setting
Acronym: MADESIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Université Libre de Bruxelles (Other); Fondation Kisane (Unknown); Les Amis de l'Institut (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3020
Record Dates: First submitted 2020-09-29; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-07

CONDITIONS: Adults; Hematological Malignancy; Oral Antineoplastic Agents
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-migrants: 53 non-migrant patients will be enrolled. "Non-migrants" will be defined as the group of native-born persons with a Belgian nationality or with a foreign nationality but with both parents native-born.
  Interventions: Behavioral: Measure adherence behaviors
- Migrants: 60 migrant patients will be enrolled. This group will include both "First Generation (FG) migrants" defined as the group of foreign-born persons and "Second Generation (SG) migrants" defined as people native-born but with either a foreign nationality or with one or both parents foreign-born.
  Interventions: Behavioral: Measure adherence behaviors

INTERVENTIONS:
Behavioral: Measure adherence behaviors — Conducted in the ambulatory setting of two Brussels hospitals, the MADESIO mixed-method study design combine sequentially a first quantitative explorative questionnaire-based study with a second in depth qualitative approach.
  The first 4 visits questionnaire-based survey prospectively measures adherence to OAMs and identify associated risk factors in the two sub-groups of ambulatory patients with various haematological malignancies. A combination of validated self-reported measures able to measure medication taking behaviours, assess both intentional and unintentional adherence, identify associated risk factors was selected.
  The second qualitative phase, based on the McGill Illness narrative interview design, deeper address patients' therapeutic adherence and subjective meanings.
  Other Names: Identify risk factors associated with poor-adherence in each subgroup of non-migrants and migrants; Explain any observed differences in adherence rates or associated risk factors between the two subgroups

SUMMARY:
Patients with haematologic malignancies are increasingly treated by Oral Anticancer Medications (OAMs), increasing the challenge of ensuring optimal adherence to treatment. However, except for Chronic Myelogenous Leukemia (CML) or Acute Lymphoid Leukemia (ALL), the extent of non-adherence has rarely been investigated in an outpatient setting. In Belgium, the only available data suffers from critical underrepresentation of patients from minority diverse population. In the context of increasing migration, the identification of differences in access and drug use that may lead to health disparities is crucial. Based on a sequential mixed method study design, our objectives are to measure adherence to OAMs in two subgroups of non-migrants and migrants with various haematological malignancies, to identify the associated risk factors and to explore the representations that come into play with regards to illness and adherence behaviors. Essentially, the MADESIO protocol will contribute to assess whether and why patients with migrant backgrounds are a risk group regarding adherence to OAMs.

DETAILED DESCRIPTION:
INTRODUCTION

For some years, the use of OAMs is increasing and oncological teams must deal with the challenge of ensuring optimal adherence to prescribed treatments. It has been demonstrated that poor adherence impacts the quality of response and risk of relapse. However, data are scarce regarding how cancer patients adhere to their medication plan, particularly those with malignancies other than breast cancer. Moreover, oncohaematology appears to be the poor cousin to the cancer adherence studies. Except for CML or ALL, the extent of non-adherence has rarely been investigated in an outpatient setting.

In Belgium, the only available data suffers from critical underrepresentation of patients from minority diverse population. This is even more restricting that, studies suggest considerable disparities and difficulties in communication between doctors and patients from different cultural and ethnic backgrounds. Considering that medication adherence is a complex interplay of predisposing factors, patients' knowledge and beliefs and patient-physician interactions, the underrepresentation of the key population of Migrants and Ethnic Minorities in adherence studies in oncology is critical.

In the context of increasing migration and emergence of novel oral therapeutics, it becomes urgent to identify potential differences in access, use and the quality of care that may lead to disparities in health outcomes. With the MADESIO Protocol, the investigators aim to fill this unmet need and to assess whether and why in oncohaematology, patients with migrant backgrounds are a risk group regarding adherence to OAMs.

OBJECTIVES

The primary objective of investigators is to measure the prevalence of medication adherence and persistence to OAMs in two subgroups of migrants and non-migrants with haematological malignancies. Additionally, in each subgroup, the study aims to identify the associated risk factors of adherence. Finallly, investigators aim to explain any observed differences between the 2 subgroups.

DESIGN

The MADESIO protocol is based on a prospective sequential mixed method study design able of tackling the challenges of studying adherence in haematology and in patients from diverse linguistic and cultural backgrounds.

Conducted in the ambulatory setting of two Brussels hospitals, the MADESIO design combines sequentially a first quantitative explorative questionnaire-based survey with a second in depth qualitative approach. The first 4 visits questionnaire-based survey prospectively measures adherence to OAMs and identify associated risk factors in two sub-groups of 60 migrant and 53 non-migrant ambulatory patients with various haematological malignancies. The second qualitative semi-structured interviews deeper address patients' therapeutic adherence and subjective meanings.

CLINICAL SETTING

The Institut Jules Bordet and the Centre Hospitalier Universitaire Saint-Pierre are two nearby hospitals. Located in the hearth of Brussels, their oncohaematological outpatient settings offer an ideal setting to explore the topic of migrants' adherence in the context of interethnic or intercultural medical consultations.

STUDY POPULATION

Eligible patients are adult patients with an haematological malignancy, having taken at least one OAM since minimum 30 days and having a minimum of 6 months life expectancy.

The sub-group of migrants is composed of "First Generation (FG)" migrants - the group of foreign-born persons - and of "Second Generation (SG)" migrants which are people born in Belgium but with either a foreign nationality or with one or both parents foreign-born.

QUANTITATIVE APPROACH - QUESTIONNAIRE-BASED STUDY VISITS:

Each patient will answer different questionnaires across 4 visits. Over one year will be necessary to include the 113 patients and over 18 months to cover the follow-up duration.

During the first information visit, the researcher obtains patient informed consent and collects full socio-demographic, socio-economic, linguistic and migratory characteristics. All subsequent questionnaires are self-administrated.

A combination of validated self-reported measures was selected because designed to measure medication taking behaviours, assess both intentional and unintentional adherence, identify barriers and levers to adherence, not excluding contextual and socioeconomic factors, patients beliefs or patients' appraisal of the collaborative bond with its haematologist.

1/ The Beliefs and Behaviour questionnaire (BBQ); 2/ the Tool for Adherence Behaviour Screening (TABS); 3/ The Morisky Medication Adherence Scale-8 (MMAS-8), 4/ The Beliefs about Medicine Questionnaire (BMQ); 5/ the Human Connection Scale (HCS);and 6/ the Hospital Anxiety and Depression Scale (HADS) was also added to screen both anxiety and depression as they can affect adherence to medications.

The TABS and MMAS-8 aiming to measure adherence behaviour are repeated at every visit. Other selected questionnaires aiming to explore the associated risk factors are distributed across the next three visits. The schedule of the next three visits is adapted according to the usual follow-up frequency of the patient. Depending on the malignancy, patients are usually monitored every one, two or three months. Visit 2 might be on Month 1, 2 or 3, visit 3 on Month 3, 4 or 6 and visit 4 to Month 6 or 9. A last questionnaire aims to capture the trend of individuals to social desirability.

At every visit, diagnosis, disease stage, prescribed drug regimen, side effects, concomitant medications, comorbidities and performance status are collected from patient medical record. After consultation, the haematologist completes contextual information regarding the presence of family members, language(s) used in communicating, assistance of an (non)-professional interpreter, and estimates the patient's level of French proficiency and the duration of the consultation.

PATIENT SELECTION AND ENROLLMENT

The researcher has access to the consultations' planning and the patients' medical file to identify potentially eligible patients. All of them are listed and selected in running order

During an initial phone contact, the researcher briefly explains the purpose of the study. If the patient agrees, a half-hour information visit is scheduled during the next regular follow-up visit. In case of language barrier, the contact person mentioned in the patient's medical file is joined and the information visit is organized in the presence of an intercultural mediator.

Questionnaires are distributed by the researcher just after the blood test, usually scheduled one to two hours before the medical consultation. All questionnaires are pre-coded with the patient study number and visit date and given to the patient in an pre-coded study envelope. The patient can then complete the questionnaires at its best convenience during the hospital visit and slide it into one of the numerous mailbox before leaving the hospital.

TRANSLATION AND VALIDATION OF THE QUESTIONNAIRES

Already validated translated versions existed in the five target languages (French, Dutch, Arabic, Polish, Romanian) for the HADS and were obtained after the licence fees. For other non-translated questionnaires, consistent with available resources and international guidelines, the investigators established a rigorous, appropriate and user-friendly valid translation method.

Forward Translation : The initial translation from the original language has been made by a professional translator, familiar with health and medical terminologies. Instructions were given in the approach to translating, emphasizing conceptual rather than literal translations, as well as the need to use natural and acceptable language for the broadest audience.

Back Translation : Using the same approach, the instrument was then converted back to English by an independent translator whose mother tongue was English and who was not familiar with the questionnaire.

Both source-questionnaire in English and Backward translation were submitted for comparison to the main researcher. Each item of the two versions were ranked in terms of comparability of language and similarity of interpretability. All discrepancies, misunderstandings or unclear wording revealed by the back-translation were discussed with a third independent translator and again translated if needed.

Preliminary pilot testing : The researcher pilot tested the prefinal version of the translation with cognitive debriefing on, first one bilingual patient with an haematological malignancy and, second, one bilingual nurse in oncology.

All suggestions for linguistic and cultural adaptation were discussed with the researcher, the two bilingual respondents and the third professional translator until a consensus is reached.

QUALITATIVE APPROACH - McGill ILLNESS NARRATIVE INTERVIEWS(MINI):

Quantitative research methods have significant limitations in capturing the complexity of human behaviour and experience, tending to ignore the social and discursive contexts in which individual and collective understandings of illness experience emerge. Understanding the meaning that haematological cancer patients give to their illness and treatment experience may be crucial to explain the statistical associated between variables observed in quantitative study.

According to an explanatory design, MADESIO study is a two-phase mixed methods design. Qualitative data will help to explain initial quantitative results. Given the lack of previous available data the two phases will be connected at two levels. A 6 months intermediate analysis of quantitative results will, on the one hand, instruct the appropriate participants to be selected for qualitative study, and on the other hand,will focus the results that need to be examined in more details. At this stage, it cannot be said whether adherence rates or associated risk factors will be different in the migrant and non-migrant subgroups. But whatever, qualitative study aims to understand why these results differ or not.

The MINI will guide the conversation and produce narratives given access the many representations that come into play with regards to illness and health-related behaviour. Especially, addressing the discursive contexts in which individual and collective understandings of illness experience emerge may contribute to understand any potential association between personal or cultural beliefs and adherence behaviours. Therefore, the structured dimension of the MINI will enable the comparison between groups of patients from different cultural background.

Sampling the selection criteria will be designed based on the first results of the quantitative study. The research team considers selecting outliers from the regression analysis or decide to learn more about the differences between people who score either high or low on adherence variables. Considering the risk of relapse or death of cancer patients treated by oral anticancer medication, the researcher will further decide to recontact appropriate members of our original quantitative sample, or to draw a new sample that meets our purposive criteria.

CONCLUSION:

When building this protocol, investigators are aware of the complexity, if only for practical reasons, of studying prospectively adherence in patients with a language barrier. Using a mixed method approach, the MADESIO protocol is able to generate solid complementary information on adherence behaviour and associated determinants among both non-migrant and migrants patients with various haematological malignancies.

Successfully addressing the challenges raised by adherence study in haematology and in minority diverse populations, this sequential mixed method design will provide a first overview of how non-migrants and migrants with haematological malignancies, in our two Brussels Hospitals, adhere to their OAMs and will contribute to understand whether and why FG and SG migrants constitute a specific population regarding adherence to OAMs.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adult (≥ 18)
* Any diagnosis of haematological malignancy
* Treatment by minimum one OAM
* Treatment since minimum 30 days
* At least 6 months of life expectancy.
* Being able to speak and read French, Dutch, English, Polish, Romanian, or Arabic.

EXCLUSION CRITERIA:

* Illiterate patient.
* Uncontrolled acute psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-Migrant and Migrants with haematological malignancies.
  Migrant group is composed of :
  "First Generation (FG)" migrants : the group of foreign-born persons "Second Generation (SG)" migrants : the group of people born in Belgium but with either a foreign nationality or with one or both parents foreign-born.
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Medication adherence Behaviour | October 2020-October 2021
  Among the scales able to measure medication-taking behaviour, the Tool for Adherence Behaviour Screening (TABS) screens both intentional and unintentional nonadherence, but also both under and overutilization. Divided in 4 items assessing adherence and 4 assessing non-adherence, all items can be answered by a 5 point-Likert-scale scale (from 'never'=1 to 'always'=5) expressing how often patients manage pharmacological and non-pharmacological disease to ensure adherence.
  Two levels of adherence will be considered (Good adherence: Differential of ≥15 ; Suboptimal adherence: Differential of ≤14) but a continuous variable is measurable by converting TABS scores into ratios of the total score.
  This measure will be repeated at every visits.
Medication adherence Behaviour and Barriers to adherence | October 2020-October 2021
  The Morisky Medication Adherence Scale (MMAS-8) is both able to measure medication-taking behaviour and identify barriers to adherence.
  This 8 items scale can identify implementation and discontinuation and can also distinct intentional from unintentional adherence. The first seven items have a dichotomous answer (yes/no) that indicates adherent or non-adherent behaviour. For item 8, patient can choose an answer on a 5-point Likert scale, expressing how often happens that a patient does not take his medications. MMAS-8 scores can range from 0 to 8 points. Three levels of adherence may be considered (low: scores of 0 to <6; medium: 6 to <8; high: 8) but a continuous variable is measurable by converting MMAS scores into ratios of the total score. This measure will be repeated at every visits.
Beliefs and Adherence Behaviour | October 2020-October 2021
  We selected a combination of validated scales eliciting the factors identified as relevant domains of interest in the study of adherence behaviours. Among them, the Beliefs and Behaviour Questionnaire (BBQ) appears particularly relevant for a first exploration of adherence behaviours and barriers to adherence. This useful, simple, socially and culturally relevant 21 close-ended questionnaire covers the various themes of adherence in adequate depth. This questionnaire measure the patient's beliefs and experiences on 5-point-Likert type scales. The Beliefs Section has two subscales of 9 and 5 statements measuring respectively the patients' confidence in their disease management and the concerns about their disease management. Experience section has two subscales of 3 and 5 statements measuring respectively the patients' satisfaction about their management and the patients' disappointment about their management. This measure will be completed on visit 2.
Beliefs about Medicine | October 2020-October 2021
  The 18 items Beliefs about Medicine Questionnaire (BMQ) allows to quantify and compare patient's personal beliefs about the necessity of their prescribed medication and their concerns about taking it. Patients who believe their medication to be necessary and have more concerns have consistently been shown to be more adherent in a range of diseases. Beliefs about medicines that may influence adherence must therefore be screened when exploring adherence among culturally diverse population.The BMQ is composed of two scales. The BMQ-Specific assessing beliefs about the necessity and the concerns about prescribed medication. The BMQ-General assessing the background general attitudes to medicines (beliefs that medicines are harmful, addictive, poisons which should not be taken continuously and that medicines are overused by doctors) which may determine the These general the person's general orientation to the prescription. This measure will be completed on visit 2.
Therapeutic Alliance | October 2020-October 2021
  On visit 3, patient completes the Human Connection Scale (HCS) to measure its appraisal of the therapeutic alliance, i.e. the collaborative bond between her or she and its haematologist. This 16-items scale is designed to evaluate the extent to which the patient feels 1) that the oncologist listens to and understands the patient's concerns about the illness 2) that the relationship involves mutual caring and respect 3) that the patient understands the information being shared by the oncologist 4) that the patient trusts the oncologist and 5) that the oncologist and patient work well together.
  For each item, the points of each 4 point-likert-scale answer are summed to give the Human Connection Score possibly ranging from 16 to 64. A higher HCS score indicates a greater Therapeutic Alliance.
Anxiety and Depression | October 2020-October 2021
  On visit 3, patient also completes the Hospital and Anxiety Depression Scale scale (HADS). Depression, anxiety, fears or anger about the illness can bring about an adverse attitude towards therapy which can affect medication adherence. Our study will invariably enrol patients with various hemopathies and prognosis, more or less far in the lines of treatment, who experience different level of stress or anxiety. The HADS provides a simple reliable tool to screen both anxiety and depression in people with physical health problems. Divided in two scales of 7 items scoring respectively the level of anxiety and depression.
  Analysed separately, scores of each 4 point-Likert-scale answer (0-3) are summed and range from 0 to 21 for anxiety and from 0 to 21 for depression. Cut-off scores are available for each scale for quantification.
Understanding of observed difference in quantitative results between the subgroup of non-migrant and migrant patients | July 2021 - December 2021
  Understanding the meaning that haematological cancer patients give to their illness and treatment experience may be crucial to explain the statistical associated between variables observed in quantitative study. Based on the McGill Illness Narrative interview we will produce narratives that give access the many representations that come into play with regards to illness and health-related behaviour. Especially, addressing the discursive contexts in which individual and collective understandings of illness experience emerge may contribute to understand any potential association between personal or cultural beliefs and adherence behaviours.

SECONDARY OUTCOMES:
Social Desirability Bias | October 2020-October 2021
  On first visit, patient completes an auto-administrated social desirability scale. The Social desirability is usually defined as "the tendency of individuals to present themselves favorably with respect to current social norms and standard" and is considered a potential and typical bias in the measurement of self-reported adherence. By adding the Social Desirability Scale-17 (SDS-17) investigators aim to improve their ability to assess whether observed differences may be the reflection of differences in willingness to report such behaviour or beliefs.
  In the 16 items Social Desirability Scale-17 (SDS-17), compared to each statement, the patient is asked to assess if this statement describes him/her or not, answering by "true" or "false". Then points will be summed across items, ranging from 0-16. A higher SDS-17 score indicates a greater social desirability.

CONTACTS AND LOCATIONS:
Overall Officials: Fati Kirakoya, PhD, Study Director — Université Libre de Bruxelles; Sandra Tricas-Sauras, PhD, Study Director — Université Libre de Bruxelles
Locations (2):
- Belgium (2):
  - CHU Saint Pierre, Brussels
  - Institut Jules Bordet, Brussels

REFERENCES:
- [Background] 1) Noens et al. (2009). Prevalence, determinants, and outcomes of nonadherence to imatinib therapy in patients with chronic myeloid leukemia: the ADAGIO study. Blood. 113(22), 5401-11. 2) Bhatia et al. (2012). Nonadherence to Oral Mercaptopurine and Risk of Relapse in Hispanic and Non-Hispanic White Children With Acute Lymphoblastic Leukemia: A Children's Oncology Group study. J. Clin. Oncol. 30(17), 2094-101. 3) Ruddy et al. (2009) Patient adherence and persistence with oral anticancer treatment. CA: A Cancer Journal for Clinicians, 59(1):56-66 4) Greer et al. A systematic review of adherence to oral antineoplastic therapies. Oncologist 2016; 21:354-376 5) Hall et al.(2016) To adhere or not to adhere: Rates and reasons of medication adherence in haematological cancer patients, Critical Reviews in Oncology/Hematology. 97:247-262 6) Lepièce (2016). Discrimination dans la consultation médicale interethnique de médecine générale ? (PhD. Thesis), UCL. 7) Van Keer et al. (2015). Conflicts between healthcare professionals and families of a multi-ethnic patient population during critical care: an ethnographic. Critical Care. 19 (441). 8) Van Wieringen et al. (2002). Intercultural communication in general practice. European Journal of Public Health. 12, 63-68 9) Sleath et al. (2003) Hispanic ethnicity physician-patient communication, and antidepressant adherence. Compr Psychiat. 44:198-204. 10) Cooper et al. (2003) Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med, 139:907-15. 11) Nieuwkerk PT, et al. Self-reported adherence is more predictive of virological treatment response among patients with a lower tendency towards socially desirable responding. Antivir Ther. 2010;15:913-916. 12) Stöbber (2001) The Social Desirability Scale-17 (SDS-17) European Journal of Psychological Assessment, 17, pp. 222-232 13) George et al. (2005) Development and validation of the Beliefs and Behaviour Questionnaire (BBQ). Patient Education and Counseling.64(1-3): 50-60 14) Garfield et al. Suitability of measures of self-reported medication adherence for routine clinical use: a systematic review. BMC Med Res Methodol. 2011; 11:149. 15) Morisky, D. E., et al. (2008). Predictive Validity of A Medication Adherence Measure in an Outpatient Setting. Journal of Clinical Hypertension (Greenwich, Conn.), 10(5), 348-354. 16) George et al. (2005) Development and validation of the Beliefs and Behaviour Questionnaire (BBQ). Patient Education and Counseling.64(1-3): 50-60 17) Wang et al. Psychometric properties of the 8-item Morisky Medication Adherence Scale in patients taking warfarin. Thromb Haemost 2012; 108: 1-7. 18) Reynolds et al. Psychometric properties of the Osteoporosis-specific Morisky Medication Adherence Scalein postmenopausal women with osteoporosis newly treated with bisphosphonates. Ann Pharmacother 2012; 46: 659-70. 19) Horne, R., et al. Self-regulation and self-management in asthma: exploring the role of illness perceptions and treatment beliefs in explaining non-adherence to preventer medication. Psychol Health 2002; 17: 17-32. 20) Horne et al. (1999). Beliefs about medicines questionnaire (BMQ). Psychology and Health. 14:1-24. 21) Mack et al. (2009) Measuring therapeutic alliance between oncologists and patients with advanced cancer: The human Connection Scale. Cancer. 115 (14):3302-3311 22) Jing et al. Factors affecting therapeutic compliance: A review from the patient's perspective Ther Clin Risk Manag. 2008 Feb; 4(1): 269-286 23) Snaith (2003) The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 1:29. doi:10.1186/1477-7525-1-29 24) Zerbe et al. (1987). Socially desirable responding in organizational behaviour: A reconception.Academy of Management Review, 12, 250-264 25) Cha et al., Translation of scales in cross-cultural research: issues and techniques. Jan Research Methodology, 10.jan 2017, pg.386-395 26) bombardier, F. et al. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec; 46(12):1417-32. 27) Groleau et al. (2006). The McGill Illness Narrative Intervew (MINI): an interview schedule to elicit meanings and modes of reasoning related to illness experience. Transcultural Psychiatry, 43(4):671-691. 28) Weiner (1985). 'Sponteneous' causal thinking. Psychology Bulletin, 97, 74-84 29) Krousel-Wood et al. New medication adherence scale versus pharmacy fill rates in seniors with hypertension.Am J Manag Care 2009; 15: 59-66. 30) Ross et al. Patient compliance in hypertension: role of illness perceptions and treatment beliefs. J Hum Hypertens 2004; 18: 607-13 31) Berglund et al. Adherence to and beliefs in lipid-lowering medical treatments: a structural equation modeling approach including the necessity-concern framework. Patient Educ Couns 2013; 91: 105-12. 32) etc.